CLINICAL TRIAL: NCT04529239
Title: A Triple Cohort, Prospective Observational Study to Analyze Type 2 Diabetes Glucose Biomarkers With a Continuous Glucose Monitoring System
Brief Title: Type 2 Diabetes Glucose Biomarker Study With a Continuous Glucose Monitoring System
Status: Completed | Type: Observational
Sponsor: Klick Inc. (Industry)
Collaborators: Mittal Global Clinical Trial Services (Unknown)
Responsible Party: Sponsor
Other Study IDs: 036033
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2020-08

CONDITIONS: Healthy; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples to collect glycated hemoglobin (HbA1c) measurements, fasting plasma glucose (FPG), and plasma glucose during an oral glucose tolerance test (OGTT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Low to Moderate Risk: The CANRISK Canadian Diabetes Risk Questionnaire will be used for study group categorization to assess who is at risk of having prediabetes or type 2 diabetes. Participants will be categorized into one the following groups: i) low to moderate risk; ii) high risk, iii) very high risk.
  Interventions: Device: Abbott Freestyle Libre Pro
- High Risk: The CANRISK Canadian Diabetes Risk Questionnaire will be used for study group categorization to assess who is at risk of having prediabetes or type 2 diabetes. Participants will be categorized into one the following groups: i) low to moderate risk; ii) high risk, iii) very high risk.
  Interventions: Device: Abbott Freestyle Libre Pro
- Very High Risk: The CANRISK Canadian Diabetes Risk Questionnaire will be used for study group categorization to assess who is at risk of having prediabetes or type 2 diabetes. Participants will be categorized into one the following groups: i) low to moderate risk; ii) high risk, iii) very high risk.
  Interventions: Device: Abbott Freestyle Libre Pro

INTERVENTIONS:
Device: Abbott Freestyle Libre Pro — Continuous glucose monitoring device to analyze diabetes biomarkers.

SUMMARY:
Current gold standard methodologies for diagnosing type 2 diabetes (T2D) or prediabetes can be unreliable and inaccurate, and require the need for multiple different tests for comparison. It is possible that a simpler and more refined method of diagnosing T2D or prediabetes involves examining the proportional-integral (PI) control system of the body's glycemic function (i.e., a model of the glucose curve). The purpose of this research is to examine how well a PI model can diagnose nondiabetic, prediabetic, or diabetic patients based on glucose data gathered from a wearable glucose monitoring device.

ELIGIBILITY:
Inclusion Criteria:

* Either male or non-pregnant, non-lactating female aged > 18-60 <years (both inclusive)
* Subjects willing to give written informed consent
* Healthy Volunteers
* Subjects able to comply with the study protocol
* Women of child bearing potential must have a negative urine pregnancy test prior to study entry
* Minimum 4 subjects in each interval of approx 7 years (18-25/26-32/32-38/39-45/46-52/53-59)
* Minimum 40% subjects of one gender to mark relative distribution

Exclusion Criteria:

* Any person below the age of 18 years
* Suspected or confirmed pregnancy
* Currently breastfeeding
* Diagnosis of any known chronic or acute medical disease of any kind (e.g., cardiovascular disease, respiratory disease, influenza, pneumonia, etc.)
* Diagnosis of any known neurological disease or psychological disorder of any kind (e.g., brain lesion, epilepsy, anxiety, eating disorder, mood disorder, sleep disorder, etc.)
* Any implanted electrical medical device (e.g., pacemaker, insulin pump, deep brain stimulator, etc.)
* Any form of prescription medication
* Use of antibiotics in the three months prior to enrollment
* Any person planning to undergo a Magnetic Resonance Imaging (MRI), Computed Tomography (CT) scan, or high-frequency electrical heat (diathermy) treatment during the duration of the study (as per restrictions of the FreeStyle Libre pro device)

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Healthy adults and those at risk of developing prediabetes or type 2 diabetes.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Glucose biomarker data from the continuous glucose monitoring device, which will be analyzed as a function of different homeostasis responses from the 3 different cohorts of individuals (i.e., i) low to moderate risk; ii) high risk, iii) very high risk). | The device is worn for 14 days on each participant
  Continuous glucose data from the FreeStyle Libre device will be collected from each individual and analyzed for differences in glucose responses (i.e., "ups" and "downs") across the different study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Klick Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaufman JM, van Veen L, Fossat Y. Screening for Impaired Glucose Homeostasis: A Novel Metric of Glycemic Control. Mayo Clin Proc Digit Health. 2023 May 24;1(2):189-200. doi: 10.1016/j.mcpdig.2023.02.008. eCollection 2023 Jun. PMID 40206722